CLINICAL TRIAL: NCT02263443
Title: Appropriated Bowel Preparation Before Exploratory Laparotomy in Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Collaborators: Prapaporn Suprasert (Unknown)
Responsible Party: Principal Investigator, Wasakorn Suadee, M.D., Chiang Mai University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: OBG-2557-02203
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Cathartic Colon; Other Surgical Procedures
Keywords: bowel preparation; gynecologic surgery; laparotomy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Soap sus enema (S.S.E.) (Experimental): Patients in S.S.E. group will receive bowel preparation by soap suds enema until clear at night before surgery.
  Interventions: Procedure: Soap suds enema (S.S.E.)
- sodium chloride enema (Experimental): Patients in unison enema group will receive Unison enema 100 ml per rectal at night before surgery.
  Interventions: Procedure: sodium chloride enema
- no enema (Placebo Comparator): Patients will receive none of bowel preparation. NPO after midnight
  Interventions: Procedure: No enema

INTERVENTIONS:
Procedure: Soap suds enema (S.S.E.) — Patients in S.S.E. group will bowel preparation by soap suds enema until clear at night before surgery.
  Arms: Soap sus enema (S.S.E.)
Procedure: sodium chloride enema — Patients in unison enema group will Unison enema 100 ml per rectal at night before surgery
  Arms: sodium chloride enema
Procedure: No enema — Patients NPO groups will NPO and no bowel preparation.
  Arms: no enema

SUMMARY:
Our study perform In Department of Gynecology, Faculty of Medicine, Chiang Mai University. In our study we divide patients into 3 groups ,First group patients doing Soap suds enema (S.S.E.), second group patients doing sodium chloride enema and the last group patient Non per os (NPO) before surgery. Our hypothesis is no different about surgical view in 3 groups and lower side effects in patients in no bowel preparation group.

Research objectives

1. Comparing the surgeon satisfaction ,surgical view and bowel handling in operation of soap suds enema group, sodium chloride enema group and the NPO group in patients under going exploratory laparotomy in gynecologic surgery.
2. Comparing the side effects of soap suds enema group, sodium chloride enema group and the NPO group.

Inclusion Criteria

1. Women under going laparotomy in gynecologic surgery 2. Surgeon consider not too difficult surgery. 3. Can understanding Thai language. 4. Can communicate with researcher. 5. Consenting participants. Exclusion Criteria

1. Pregnancy or suspected pregnancy.
2. Laparoscopic surgery
3. Do not consent to participate in research
4. Gastrointestinal infection
5. Underlying disease such as Intestinal disease, patient who cannot under going bowel preparation ,heart disease ,seizure.
6. Surgeon consider difficult surgery such as fixed mass or uterus with others organs from per vaginal examination or very huge mass or history of difficult surgery or history of severe adhesion in abdominal cavity.

DETAILED DESCRIPTION:
Methods

1. Divide patients into 3 groups ,First group patients doing Soap suds enema (S.S.E.), second group patients doing sodium chloride enema and the last group patient Non per os (NPO) before surgery
2. Patients information such as age, height, weight, smoking, history of surgery, number of surgeries, diagnosis that required surgery. The complete blood count and the laboratory prior to surgery record by the research team.
3. Patients do self questionnaire about symptoms such as abdominal pain or discomfort , anxiety ,nausea and vomiting etc. these are for understanding symptoms of patients before bowel preparation perform.
4. Computer-generated sequence into block for 30 person
5. Random into 3 groups by nurses .in opaque envelopes with number infront of to identify patients. Surgeon must not know what group of these patients get in.
6. Patients in S.S.E. group will bowel preparation by soap suds enema until clear at night before surgery.
7. Patients in unison enema group will Unison enema 100 ml per rectal at night before surgery
8. Patients NPO groups will NPO and no bowel preparation.
9. Patients in all group are doing operative preparation such as NPO after midnight, retained foley catheter and clean abdomen and perineum before surgery. Closs matching blood.
10. In the morning before surgery , patients do self questionnaire about symptoms score such as abdominal pain or discomfort , anxiety ,nausea and vomiting etc. for symptoms of patients after bowel preparation perform last night.
11. In operation room , surgeon evaluate surgical view, bowel handling after use swabs for bowel packing and record by nurse and after operation finish surgeon evaluate satisfaction of operation.
12. One day after surgery and before discharge from hospital patients do self questionnaire about symptoms score such as abdominal pain or discomfort , anxiety ,nausea and vomiting etc

ELIGIBILITY:
Inclusion Criteria:

1. Women under going laparotomy in gynecologic surgery
2. Surgeon consider not too difficult surgery.
3. Can understanding Thai language.
4. Can communicate with researcher.
5. Consenting participants.

Exclusion Criteria:

1. Pregnancy or suspected pregnancy.
2. Laparoscopic surgery
3. Do not consent to participate in research
4. Gastrointestinal infection
5. Underlying disease such as Intestinal disease, patient who cannot under going bowel preparation ,heart disease ,seizure.
6. Surgeon consider difficult surgery such as fixed mass or uterus with others organs from per vaginal examination or very huge mass or history of difficult surgery or history of severe adhesion in abdominal cavity.

Max Age: 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
surgical view and bowel handling in operation | 1 day after bowel preparation
  surgeon evaluate surgical view, bowel handling after use swabs for bowel packing and record by nurse and after operation finish surgeon evaluate satisfaction of operation.
  Evaluation in operation
  1. In operation room , surgeon evaluate surgical view, bowel handling after use swabs for bowel packing and record by nurse using visual analog scale score 0 to 10 that depend on surgical view and bowel handling, 0 is the worst surgical view and hardest bowel handling and 10 for extremely good surgical view and easiest bowel handling.
  2. When the operation finished surgeon evaluate satisfaction of operation .
Comparing the side effects of soap suds enema group, sodium chloride enema group and the NPO group. | 1 day before surgery and 3 day after surgery
  Patients self answers Questionnaire about symptoms by visual analog scale score 0 to 10 that depend on severity of symptoms 0 is no symptoms and 10 most severe symptoms.
  Symptoms including headache, nausea, vomiting, thirsty, fatique, anxious, discomfort, abdominal pain , bloating, insomnia, ashamed, fecal incontinence.
  Additional questions in morning before surgery are Do you feelng discomfort from these bowel preparation?, do you want to do the same bowel preparation method if you have to do next operation? and do you want to change to other methods?,

CONTACTS AND LOCATIONS:
Overall Officials: Prapaporn - Suprasert, Study Director — Chiang Mai University
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine, Chiang Mai University, Amphoe Muang, Chiang Mai, Thailand